CLINICAL TRIAL: NCT04462809
Title: A Three-Cohort Phase II Trial to Assess the Efficacy of a Maintenance Treatment With TALAzoparib Following First Line Platinum-based Chemotherapy in Pleural or Malignant Peritoneal MESOthelioma Patients
Brief Title: Efficacy of a Maintenance Treatment With TALAzoparib Following First Line Platinum-based Chemotherapy in Malignant MESOthelioma
Acronym: TALAMESO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL19_0457
Record Dates: First submitted 2020-07-06; First posted 2020-07-08 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Advanced Malignant Pleural or Peritoneal Mesothelioma
Keywords: Talazoparib; maintenance-based treatment; PARP-inhibitor; malignant pleural mesothelioma; malignant peritoneal mesothelioma; predictive biomarkers
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — talazoparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A, Malignant pleural mesothelioma (Experimental): Malignant pleural mesothelioma
  Interventions: Drug: Talazoparib
- Cohort B1:Malignant peritoneal mesothelioma non-resected (Experimental): Malignant peritoneal mesothelioma with non-resected or incompletely resected disease
  Interventions: Drug: Talazoparib
- Cohort B2:Malignant peritoneal mesothelioma (resected) (Experimental): Malignant peritoneal mesothelioma with completely resected disease.
  Interventions: Drug: Talazoparib

INTERVENTIONS:
Drug: Talazoparib — Talazoparib 1 mg a day (PO) (or 0.75 mg a day) for 2 years, started between 6 to 8 weeks after the end of chemotherapy discontinuation.
  Talazoparib will be given for up to 2 years, or less length of time in the case of disease progression,.
  unacceptable toxicity despite adequate management,patient decides to withdraw from the study, or general or specific changes in the patient's condition render the patient unacceptable for further treatment.

SUMMARY:
Malignant mesothelioma is an invasive neoplasm that arises from mesothelium that lines several organs. Common primary sites of origin of mesotheliomas are the pleura (malignant pleural mesothelioma: 85%) and peritoneum (malignant peritoneal mesothelioma 15%), and rarely the pericardium and tunica vaginalis.

The standard of care recommended for malignant pleural mesotheliomas (MPM) is palliative chemotherapy based on a doublet of platinum salt and an anti-folate. The median survival of patients with pleural MPM is around 8 months with best supportive care only, 12 to 19 months when systemic chemotherapy is used with or without anti-angiogenic agents or targeted therapy. There is an unmet need for innovative approaches in pleural mesotheliomas.

Malignant peritoneal mesothelioma is an aggressive neoplasm that arises from the lining mesothelial cells of the peritoneum and spreads extensively within the confines of the abdominal cavity. Cytoreductive surgery (CRS) followed by hyperthermic intraoperative peritoneal perfusion with chemotherapy (HIPEC) is the standard curative approach when it is possible, with respect to peritoneal carcinomatosis extend. When the cytoreductive surgery is impossible, the common strategy is to prescribe systemic chemotherapy, with the objective of downsizing tumor lesions for potential subsequent CRS. The standard strategy based on cisplatin - pemetrexed combination regimen has been extrapolated from pleural mesothelioma management principles.

Genomic landscape of mesotheliomas is now well described. Pleural and peritoneal malignant mesotheliomas harbor closed genomic instability.

Strategies based on maintenance-based treatments with Poly (ADP-ribose) polymerase (PARP) inhibitors, especially olaparib, niraparib and talazoparib, have been shown effective in ovarian cancer patients, thereby leading to their approvals. The benefit has been mainly observed in patients with homologous recombination deficiencies (HRD), but also in all-comers patients in a lesser extent. It is thought that HRD induces addiction of cancer cells to PARP, thereby leading to cell death in the presence of PARP inhibitors.

As a consequence, given the prevalence of HRD, through BAP-1 mainly, in mesotheliomas, maintenance treatment with PARP-inhibitor in malignant mesothelioma patients without any progressive disease after 4 to 6 cycles of platinum-based chemotherapy may be associated with increased progression free survival, as it was shown in ovarian cancer patients.

TALAMESO aims to evaluate the efficacy of talazoparib maintenance treatment given for maximum 2 years following 4 to 6 cycles of platinum-based first line chemotherapy in terms of proportion of patients progression free 6 months after starting the maintenance, and progression-free survival, in patients with advanced malignant pleural (cohort A) or peritoneal (cohorts B1 and B2) mesotheliomas.

Cohorts B1 and B2 are meant to confirm that talazoparib can increase progression free survival in both patient populations with non-resected or incompletely resected disease (cohort B1) or with completely resected disease (cohort B2).

TALAMESO is an open-label phase II trial with 3 independent cohorts (Fleming's single-stage) including patients with advanced malignant pleural (cohort A) or peritoneal (cohort B1 and B2) mesotheliomas without any sign of disease progression after 4 to 6 cycles of platinum-based chemotherapy (including minimum 1 cycle of pemetrexed).

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old
* Patients with Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Histologically - or cytologically - confirmed malignant mesotheliomas: epithelioid, sarcomatoid, biphasic
* Developed from pleura (cohort A) or from peritoneum (cohorts B1 and B2)
* Previously treated with first-line platinum based-chemotherapy (including minimum one cycle of pemetrexed) for 4 to 6 cycles, with no sign of disease progression during chemotherapy.
* No previous treatment with bevacizumab and PARP inhibitor
* Minimum 6 weeks and maximum 8 weeks interval between last chemotherapy cycle and talazoparib start
* For pleural mesotheliomas (cohort A), primary or interval debulking surgery with or without hyperthermic intrapleural or intrathoracic chemotherapy (HITHOC) will be authorized, in the case of non-complete cytoreductive surgery only
* For peritoneal mesotheliomas

  * In cohort B1, primary or interval debulking surgery ± hyperthermic intraperitoneal chemotherapy (HIPEC) will be authorized in the case of non-complete cytoreductive surgery (CC2 or CC3) only. This cohort will also include patients with non-operated diseases
  * In cohort B2, complete macroscopic (CC0 or CC1) primary or interval debulking surgery ± HIPEC will be required.

Intraperitoneal treatment with pressurized intraperitoneal aerosol chemotherapy sessions (PIPAC) are not allowed.

* Measurable or non-measurable (but radiologically evaluable) disease as per modified RECIST version 1.1 on computed tomography (CT) scan (within 28 days of talazoparib initiation)
* Availability at the study site of a representative FFPE tumor sample in a block or at least 30 unstained slides from biopsy or surgery specimen, aged less than 6 months.
* Patients with adequate bone marrow function measured within 28 days prior to administration of study treatment as defined below:
* Absolute neutrophil count ≥1.0 x 109 /L
* Platelet count ≥50 x 109 /L
* Haemoglobin ≥8.0 g/dL (may have been blood transfused)
* Patients with adequate renal function:
* Calculated Glomerular Filtration Rate (GFR) ≥30 ml/min/1.73 m2 according to CKD-EPI formula
* Patients with adequate hepatic function
* Total bilirubin ≤ 1 × upper limit of normal [ULN] and aspartate aminotransferase (AST) > ULN
* Total bilirubin > 1.0 to1.5 × ULN and any AST
* Patients must have a life expectancy ≥16 week.
* Confirmation of non-childbearing status (pregnancy test) for women of childbearing potential.
* A highly effective method of contraception is required for female patients during treatment of talazoparib, and for at least 7 months after completing therapy. Advise male patients with female partners of reproductive potential and pregnant partners to use a condom, during treatment with talazoparib and for at least 4 months after the final dose.
* Patients who gave its written informed consent to participate to the study.
* Patients affiliated to a social insurance regime.
* Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

* Uncontrolled intercurrent illness, including but not limited to, such as congestive heart failure; respiratory distress; liver failure; allergy, or psychiatric illness/social situations that would limit compliance with study requirement according to the investigator, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
* Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≥5 years.
* All subjects with brain metastases or meningeal involvement.
* Patients receiving any systemic chemotherapy, radiotherapy (except for palliative reasons), within 6 weeks from the last dose prior to study treatment (or a longer period depending on the defined characteristics of the agents used). The patient can receive a stable dose of bisphosphonates for bone metastases, before and during the study as long as these were started at least 4 weeks prior to treatment with study drug.
* Persistent toxicities (CTCAE ≥grade 2) with the exception of alopecia and sensory neuropathy, caused by previous cancer therapy.
* Treatment with other investigational agents.
* Bowel occlusive syndrome, inflammatory bowel disease, immune colitis, or other gastro-intestinal disorder that does not allow oral medication such as malabsorption.
* Known severe hypersensitivity reactions to PARP inhibitors.
* Known HIV or AIDS related illness.
* Positive test for HBV surface antigen and / or confirmatory HCV RNA (if anti-HCV antibody tested positive).
* Treatment with oral anticoagulant anti-vitamin K such Coumadin®
* Prior organ transplantation, including allogeneic stem cell transplantation (excluding autologous bone marrow transplant).
* Patients under guardianship.
* Women who are breastfeeding (during treatment with talazoparib and for at least 1 month after the final dose)
* Participation in other interventional clinical research that may interfere with the experimental drugs efficacy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Non-progression proportion | 6 month after starting talazoparib
  The non-progression proportion is defined as the proportion of patients free of progression 6 months after talazoparib start. Disease progression will be based on (i) tumor assessment made by the investigators according to the RECIST 1.1 criteria and/or, ii) non-equivocal clinical symptom of disease progression according to the investigator; (iii) death related to disease progression.

SECONDARY OUTCOMES:
Progression free survival | Patients will be followed until the end of the study for collect date on progression and date of eventually death : .25 month for the latest enrolled patient to 49 months for the first one.)
  The Progression-Free Survival (PFS) is defined as the time from inclusion to (1) first documented disease progression or death related to disease progression, whichever occurs first or, (2) end of follow-up.
Progression free-survival based on RECIST 1.1 criteria | Patients will be followed until the end of the study for collect date on progression and date of eventually death : .25 month for the latest enrolled patient to 49 months for the first one.
  The Progression-Free Survival (PFS) is defined as the time from inclusion to first documented disease progression or death related to disease progression, whichever occurs first or, end of follow-up. Disease progression will be based on tumor assessment made by the investigators according to the RECIST 1.1 criteria and/or, non-equivocal clinical symptom of disease progression according to the investigator, and/or death related to disease progression.
Progression free-survival based on mRECIST criteria | Patients will be followed until the end of the study for collect date on progression and date of eventually death : .25 month for the latest enrolled patient to 49 months for the first one.
  The Progression-Free Survival (PFS) is defined as the time from inclusion to first documented disease progression or death related to disease progression, whichever occurs first or, end of follow-up. Disease progression will be based on tumor assessment made by the investigators according to the mRECIST criteria and/or, non-equivocal clinical symptom of disease progression according to the investigator, and/or death related to disease progression.
Overall Survival | Patients will be followed until the end of the study for collect date on progression and date of eventually death : .25 month for the latest enrolled patient to 49 months for the first one.
  The Overall Survival (OS) will be estimated from the date of inclusion to the date of death or to the end of follow-up.
Safety, treatment-related adverse events | 6 weeks after the last experimental treatment for the latest enrolled patient
  treatment-related adverse events are defined as the nature, number and grade of adverse events observed throughout the study and assessed using NCI-CTCAE v.5.0 criteria.